CLINICAL TRIAL: NCT05633264
Title: Deucravacitinib Post-marketing Surveillance in Patients With Psoriasis in Japan
Brief Title: A Study to Assess Deucravacitinib Post-marketing Surveillance in Participants With Psoriasis in Japan
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: IM011-226
Record Dates: First submitted 2022-11-22; First posted 2022-12-01 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Psoriasis
Keywords: Psoriasis; Deucravacitinib
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort 1: Psoriasis (PsO) participants who initiate treatment with Deucravacitinib.

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of deucravacitinib for the treatment of plaque psoriasis (PsO) in Japan participants.

ELIGIBILITY:
Inclusion Criteria:

* Psoriasis (PsO) participants who received Deucravacitinib for the first time of the approved indications at medical institutions in Japan will be enrolled in this PMS

Exclusion Criteria:

* Participants receiving Deucravacitinib for an off-label indication will be excluded from this PMS.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of Psoriasis (PsO) participants (participants with plaque psoriasis, generalized pustular psoriasis, and erythrodermic psoriasis) who initiate treatment with Deucravacitinib will be enrolled. Participants receiving Deucravacitinib for an off label indication will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 369 (Actual)
Dates: Start 2022-12-05 (Actual); Primary Completion 2025-05-28 (Actual); Study Completion 2025-05-28 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) | Up to 52 weeks

SECONDARY OUTCOMES:
Proportion of participants achieving Static Physicians Global Assessment (sPGA) of 0/1 during study period | Up to 52 weeks
Change from Baseline in Body Surface Area (BSA) during study period | Up to 52 weeks
Proportion of participants achieving Global Improvement Score (GIS) during study period | Up to 52 weeks
Distribution of demographic characteristics: Age | Up to 52 weeks
Distribution of demographic characteristics: Sex | Up to 52 weeks
Distribution of demographic characteristics: Height | Up to 52 weeks
Distribution of demographic characteristics: Weight | Up to 52 weeks
Distribution of demographic characteristics: Past history /complication | Up to 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- EP Pharmaline, Tosima-ku, Tokyo, Japan

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html